CLINICAL TRIAL: NCT03373461
Title: An Adaptive Seamless Randomized, Double-blind, Placebo-controlled, Dose Ranging Study to Investigate the Efficacy and Safety of LNP023 in Primary IgA Nephropathy Patients
Brief Title: Study of Safety and Efficacy of LNP023 in Patients With Kidney Disease Caused by Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNP023X2203; 2017-000891-27 (EudraCT Number)
Record Dates: First submitted 2017-11-30; First posted 2017-12-14 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: IgA Nephropathy
Keywords: glomerunephritis, complement driven, chronic kidney disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo identical to LNP023 twice a day
  Interventions: Other: Placebo
- LNP023 10 mg BID (Experimental): 10 mg taken twice a day.
  Interventions: Drug: LNP023
- LNP023 50 mg BID (Experimental): 50 mg taken twice a day.
  Interventions: Drug: LNP023
- LNP023 100 mg BID - Part 2 (Experimental): 100 mg taken twice a day.
  Interventions: Drug: LNP023
- LNP023 200 mg BID (Experimental): 200 mg taken twice a day.
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — LNP023 5, 25, 100 mg capsles
  Arms: LNP023 10 mg BID; LNP023 100 mg BID - Part 2; LNP023 200 mg BID; LNP023 50 mg BID
Other: Placebo — Matching placebo to LNP023
  Arms: Placebo

SUMMARY:
Efficacy and safety of LNP023 in IgAN patients

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, dose-ranging, parallel-group study with an adaptive design (Part 1 informed the design adaptations for Part 2). In Part 1, three doses of LNP023 (10 mg, 50 mg, and 200 mg) vs. placebo control were compared; In Part 2, four doses of LNP023 (10 mg, 50 mg, 100 mg, and 200 mg) vs. placebo control were compared. The study comprised a run-in phase in order that patients were on stable and maximally tolerated dose of Angiotensin-converting-enzyme inhibitor (ACEi) or Angiotensin II Receptor Blockers (ARB) for at least 90 days, a 90 days treatment phase in Part 1; a 180 days treatment phase in Part 2 and a 90 days follow-up phase in both Parts 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients above 18 years of age with a biopsy-verified IgA nephropathy and where the biopsy was performed within the prior three years.
* Patients must weigh at least 35 kg to participate in the study, and must have a body mass index (BMI) within the range of 15 - 38 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* Measured Glomerular Filtration Rate (GFR) or estimated GFR (using the CKD-EPI formula) ≥30 mL/min per 1.73 m2
* Urine protein ≥1 g/24hr at screening and ≥0.75 g / 24h after the run- in period
* Vaccination against Neisseria meningitidis types A, C, Y and W-135 is required at least 30 days prior to first dosing with LNP023. Vaccination against N. meningitidis type B, S. pneumoniae and H. influenzae should be conducted if available and acceptable by local regulations, at least 30 days prior to first dosing with LNP023
* All patients must have been on supportive care including a maximally tolerated dose of ACEi or ARB therapy for the individual, antihypertensive therapy or diuretics for at least 90 days before dosing

Exclusion criteria

1. Presence of crescent formation in ≥50% of glomeruli assessed on renal biopsy
2. Patients previously treated with immunosuppressive agents such as cyclophosphamide or mycophenolate mofetil (MMF), or cyclosporine, systemic corticosteroids exposure within 90 days prior to start of LNP023/Placebo dosing
3. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations
4. All transplanted patients (any organ, including bone marrow)
5. History of immunodeficiency diseases, or a positive HIV (ELISA and Western blot) test result.

   Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV). A positive HBV surface antigen (HBsAg) test, or if standard local practice, a positive HBV core antigen test, excludes a patient. Patients with a positive HCV antibody test should have HCV RNA levels measured. Subjects with positive (detectable) HCV RNA should be excluded
6. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:

   * A history of invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus
   * Splenectomy
   * Inflammatory bowel disease, peptic ulcers, severe gastrointestinal disorder including rectal bleeding;
   * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
   * Pancreatic injury or pancreatitis;
   * Liver disease or liver injury as indicated by abnormal liver function tests. ALT (SGPT), AST (SGOT), GGT, alkaline phosphatase and serum bilirubin will be tested.
   * Any single parameter of ALT, AST, GGT, alkaline phosphatase or serum bilirubin must not exceed 3 x upper limit of normal (ULN)
   * PT/INR must be within the reference range of normal individuals
   * Evidence of urinary obstruction or difficulty in voiding any urinary tract disorder other than IgNA that is associated with hematuria at screening and before dosing; [If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to randomization, to rule out any laboratory error]
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
8. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening or baseline:

   * PR > 200 msec
   * QRS complex > 120 msec
   * QTcF > 450 msec (males)
   * QTcF > 460 msec (females)
   * History of familial long QT syndrome or known family history of Torsades de Pointes
   * Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of the study
9. History of severe allergic reactions as per Investigator decision
10. Plasma donation (> 200mL) within 30 days prior to first dosing.
11. Donation or loss of 400 mL or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after stopping of investigational drug. Highly effective contraception methods include:

    * Total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure <1%), for example hormone vaginal ring or transdermal hormone contraception In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.

    If local regulations deviate from the contraception methods listed above and require more extensive measures to prevent pregnancy, local regulations apply and will be described in the ICF.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
13. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
14. History of any porphyria metabolic disorder
15. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening and baseline.
16. History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- Argentina (2):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (3):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Roeselare
- Brazil (2):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Barranquilla, Colombia
- Novartis Investigative Site, Prague, Czechia
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Arhus N
- Novartis Investigative Site, HUS, Finland, Finland
- Novartis Investigative Site, Montpellier, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- India (2):
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, New Delhi
- Israel (3):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Japan (5):
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Novartis Investigative Site, Groningen, Netherlands
- Norway (3):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Loerenskog
  - Novartis Investigative Site, Oslo
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Sweden (2):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Taiwan (3):
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (5):
  - Novartis Investigative Site, Cambridge, Cambrigdeshire
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 99 participants screened and 46 randomized participants completed in Part 1. There were 162 screened in Part 2 and 66 were randomized. All participants completed a run-in period of at least 30 days. Participants randomized to Part 1 could not participate in Part 2.
Groups:
- LNP023 100 mg BID - Part 2: 100 mg taken orally twice a day
- Placebo: Placebo identical to LNP023 taken orally twice a day
Period: Part 1
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Started | 9 | 8 | 0 | 15 | 14
Completed | 9 | 8 | 0 | 15 | 14
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Started | 11 | 11 | 22 | 11 | 11
Completed | 11 | 10 | 22 | 11 | 10
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 22 | 26 | 25 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.42) | 36.6 (8.42) | 36.0 (13.15) | 42.5 (15.76) | 39.4 (11.00) | 38.9 (12.58)
Age, Customized [Count of Participants; unit: Participants]
  18 years - <65 years | 20 | 19 | 21 | 24 | 25 | 109
  65 years - <85 years | 0 | 0 | 1 | 2 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 11 | 11 | 7 | 46
  Male | 9 | 13 | 11 | 15 | 18 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 9 | 12 | 12 | 11 | 54
  White | 10 | 9 | 10 | 13 | 13 | 55
  Black or African American | 0 | 1 | 0 | 1 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
Urine Protein to Creatinine Ratio (UPCR) [Mean (Standard Deviation); unit: g/mol] — From 24 hour urine collection
  g/mol | 214.1 (122.29) | 188.2 (90.38) | 203.4 (98.29) | 151.0 (109.46) | 146.6 (61.62) | 177.9 (100.02)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 66.0 (28.51) | 53.8 (22.73) | 67.0 (31.75) | 57.9 (28.92) | 65.7 (32.60) | 62.2 (29.30)
Supine Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Blood pressure measurements not available for all participants
  mmHg
    Systolic: number analyzed (Participants) | 12 | 12 | 11 | 18 | 17 | 70
    Systolic | 134.4 (11.65) | 122.6 (12.15) | 125.0 (11.30) | 125.7 (11.66) | 125.5 (11.37) | 126.5 (11.89)
    Diastolic: number analyzed (Participants) | 12 | 12 | 11 | 18 | 17 | 70
    Diastolic | 84.1 (7.65) | 76.9 (8.41) | 80.0 (10.40) | 79.7 (7.62) | 78.2 (7.32) | 79.6 (8.26)
Prior use of ACEi and/or ARB [Count of Participants; unit: Participants] — Prior use of angiotensin converting enzyme inhibitor and/or angiotensin receptor blocker
  Participants | 19 | 19 | 22 | 26 | 25 | 111

OUTCOME MEASURES:

1. Primary Outcome: MCP-Mod Estimates of the Ratio to Baseline of Urine Protein to Creatinine Ratio (UPCR) (g/Mol) - Parts 1 and 2 at Day 90
Description: The primary analysis of the dose-response effect of LNP023 versus placebo on the reduction in UPCR 24 hours at Day 90 was done using Multiple Comparison Procedure Modelling (MCP-Mod). The existence of a dose-response relationship was assessed at the MCP step at the one-sided 10% significance level vis a multiple contrasts test. In the Mod step, the mean predicted difference between each LNP023 dose and placebo were then estimated using parametric bootstrap model averaging. Results are presented on the original scale as geometric mean ratios. A ratio less than 1 indicates a reduction in proteinuria. Participants collected all urine over a 24 hour period for UPCR test.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 22 | 26 | 25
Ratio to baseline | 0.85 [0.77 to 0.93] | 0.80 [0.73 to 0.87] | 0.76 [0.70 to 0.81] | 0.69 [0.61 to 0.77] | 0.88 [0.80 to 1.00]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs LNP023 50 mg BID vs LNP023 100 mg BID - Part 2 vs LNP023 200 mg BID vs Placebo; Test type: Other; p = 0.038, Multiple Comparison Procedure-Modeling
Statistical Analysis 2: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.99, 80% CI 2-sided [0.86 to 1.00]
Statistical Analysis 3: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.94, 80% CI 2-sided [0.76 to 0.98]
Statistical Analysis 4: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.87, 80% CI 2-sided [0.72 to 0.96]
Statistical Analysis 5: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.77, 80% CI 2-sided [0.66 to 0.92]

2. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Change From Baseline for Estimated Glomerular Filtration Rate (eGFR) - Parts 1 and 2 at Day 90
Description: eGFR was calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI). The CKD-EPI equation is an established, widely used and Kidney Disease Improving Global Outcomes (KDIGO) guideline recommended method of GFR estimation based on serum creatinine, age, gender and race of the patient. It was derived and validated established from a meta-analyses of multiple studies including large number of patients.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: mL/min/SSA
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 20 | 19 | 22 | 26 | 25
mL/min/SSA | -0.06 (1.760) | 2.49 (1.859) | 0.23 (1.821) | 2.42 (1.545) | -3.34 (1.606)
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 3.28, 80% CI 2-sided [0.210 to 6.344]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 5.83, 80% CI 2-sided [2.642 to 9.010]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Mean Difference (Final Values) = 3.56, 80% CI 2-sided [0.427 to 6.700]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 5.76, 80% CI 2-sided [2.882 to 8.638]

3. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Change From Baseline for Serum Creatinine - Parts 1 and 2 at Day 90
Description: Serum creatinine
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 20 | 19 | 22 | 26 | 25
umol/L | -2.55 (3.488) | -2.60 (3.665) | 0.76 (3.555) | -3.47 (3.043) | 6.65 (3.150)
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = -9.20, 80% CI 2-sided [-15.253 to -3.145]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = -9.25, 80% CI 2-sided [-15.499 to -3.000]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Mean Difference (Final Values) = -5.89, 80% CI 2-sided [-12.040 to 0.260]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = -10.12, 80% CI 2-sided [-15.763 to -4.471]

4. Secondary Outcome: Shift Table From Baseline for Hematuria Levels - Parts 1 and 2 at Day 90
Description: Hematuria levels were the number of erythrocytes/high-power-field (hpf) measured through microscopic examination. The table shows the shift in hematuria grade (Low: <9 rbc/hpf, Intermediate: >=9 to <= 50 rbc/hpf, High: >50 rbc/hpf) from baseline (rows) to Day 90 (columns). A lower grade corresponds to a better outcome. Only patients with both baseline and Day 90 hematuria values are presented. L=low, I=intermediate and H=high in column headings for doses and BL=baseline
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with both baseline and Day 90 hematuria values. The number of participants analyzed corresponds to the column totals (i.e. the number of patients with non-missing baseline and day 90 values by hematuria level at Day 90 and treatment group).
Measure: Number; unit: participants
Groups:
- 10mg-L; 50mg-L; 100mg-L; 200mg-L; Pl-L: L (<9 rbc/hpf) at Day 90
- 10mg-I; 50mg-I; 100mg-I; 200mg-I; PL-I: I (>=9 to <= 50 rbc/hpf) at Day 90
- 10mg-H; 50mg-H; 100mg-H; 200mg-H; PL-H: H (>50 rbc/hpf) at Day 90
Arm/Group | 10mg-L | 10mg-I | 10mg-H | 50mg-L | 50mg-I | 50mg-H | 100mg-L | 100mg-I | 100mg-H | 200mg-L | 200mg-I | 200mg-H | Pl-L | PL-I | PL-H
Number analyzed (Participants) | 8 | 4 | 0 | 14 | 1 | 0 | 12 | 1 | 0 | 12 | 2 | 0 | 10 | 2 | 1
participants
  Low at baseline | 7 | 1 |  | 13 | 0 |  | 6 | 0 |  | 6 | 0 |  | 6 | 2 | 0
  Intermediate at baseline | 1 | 3 |  | 1 | 1 |  | 4 | 0 |  | 6 | 2 |  | 4 | 0 | 1
  High at baseline | 0 | 0 |  | 0 | 0 |  | 2 | 1 |  | 0 | 0 |  | 0 | 0 | 0

5. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline in 24hour Urine Protein (UP) - Parts 1 and 2 to Day 90
Description: Participants collected all of their urine over a 24-hour period.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 22 | 26 | 25
Ratio to baseline | 0.80 [0.661 to 0.965] | 0.89 [0.740 to 1.070] | 0.61 [0.509 to 0.729] | 0.70 [0.601 to 0.823] | 0.84 [0.713 to 0.987]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.95, 80% CI 2-sided [0.742 to 1.222]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 1.06, 80% CI 2-sided [0.830 to 1.356]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.73, 80% CI 2-sided [0.569 to 0.928]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.84, 80% CI 2-sided [0.669 to 1.050]

6. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline of 24 Hour Urine Albumin (UA) - Parts 1 and 2 to Day 90
Description: Participants collected all of their urine over a 24-hour period.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 22 | 26 | 25
Ratio to baseline | 0.79 [0.648 to 0.964] | 0.93 [0.763 to 1.122] | 0.61 [0.504 to 0.734] | 0.73 [0.623 to 0.865] | 0.82 [0.693 to 0.973]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.96, 80% CI 2-sided [0.741 to 1.250]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 1.13, 80% CI 2-sided [0.872 to 1.458]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.74, 80% CI 2-sided [0.574 to 0.957]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.89, 80% CI 2-sided [0.706 to 1.132]

7. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline in 24 Hour Urine Albumin to Creatinine (UACR) - Parts 1 and 2 to Day 90
Description: Participants collected all of their urine over a 24-hour period.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 22 | 26 | 25
Ratio to baseline | 0.85 [0.728 to 0.998] | 0.89 [0.765 to 1.045] | 0.66 [0.567 to 0.772] | 0.74 [0.647 to 0.842] | 0.87 [0.756 to 0.998]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.98, 80% CI 2-sided [0.794 to 1.214]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 1.03, 80% CI 2-sided [0.835 to 1.269]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.76, 80% CI 2-sided [0.616 to 0.942]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.85, 80% CI 2-sided [0.704 to 1.027]

8. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline in Urine Protein to Creatinine (UPCR) From 1st Morning Void - Parts 1 and 2 at Day 90
Description: A midstream urine sample was obtained from the first morning void (FMV) on the visit day.
Time Frame: Baseline and Day 90
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 20 | 19 | 22 | 26 | 25
Ratio to baseline | 0.76 [0.638 to 0.908] | 0.81 [0.674 to 0.970] | 0.61 [0.509 to 0.725] | 0.70 [0.598 to 0.815] | 0.83 [0.704 to 0.970]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.92, 80% CI 2-sided [0.723 to 1.172]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.98, 80% CI 2-sided [0.767 to 1.249]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.74, 80% CI 2-sided [0.577 to 0.937]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.84, 80% CI 2-sided [0.678 to 1.052]

9. Secondary Outcome: Plasma Pharmacokinetics (PK) of Area Under the Curve at Steady State (AUCtau,ss and AUClast,ss) at Day 30
Description: AUClast,ss: the area under the plasma concentration-time curve from time zero to last quantifiable concentration at steady state AUCtau,ss: the area under the plasma concentration-time curve from time zero to the end of the dosing interval tau at steady state
Time Frame: Baseline (0 hr), Day 15 (0 hr) Day 30 (0, 0.25, 0.5, 1, 2, 4, 6, 8 hrs)
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 18 | 18 | 16 | 24
hr*ng/mL
  AUClast,ss | 5820 (1750) | 13000 (2740) | 18400 (6040) | 27900 (9930)
  AUCtau,ss | 8010 (2550) | 17700 (4250) | 24700 (8030) | 37100 (13500)

10. Secondary Outcome: Plasma Pharmacokinetics (PK) of Pre-dose Trough at Steady State (Ctrough,ss) and Maximum Concentrations (Cmax,ss) at Day 30
Description: Cmax,ss: the observed maximum plasma concentration following drug administration at steady state (ng/mL) Ctrough,ss: the pre-dose plasma concentration observed during a dosing interval at steady state (ng/mL)
Time Frame: Baseline (0 hr), Day 15 (0 hr) Day 30 (0, 0.25, 0.5, 1, 2, 4, 6, 8 hrs)
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 18 | 18 | 16 | 24
ng/mL
  Ctrough,ss | 515 (232) | 1130 (348) | 1510 (567) | 2200 (964)
  Cmax,ss | 964 (264) | 2150 (480) | 3300 (1080) | 4940 (1770)

11. Secondary Outcome: Plasma Pharmacokinetics (PK) of Time to Maximum Concentration at Steady State (Tmax,ss) at Day 30
Description: Tmax,ss: the time to reach the maximum concentration after drug administration at steady state (h)
Time Frame: Baseline (0 hr), Day 15 (0 hr) Day 30 (0, 0.25, 0.5, 1, 2, 4, 6, 8 hrs)
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Median (Full Range); unit: hour
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 18 | 18 | 16 | 24
hour | 2.00 [0.250 to 6.00] | 2.00 [1.00 to 6.00] | 2.00 [0.500 to 6.00] | 2.00 [0.500 to 4.00]

12. Secondary Outcome: Amount of LNP023 Excreted Into Urine (Ae,ss) at Day 30
Description: Ae,ss: the total cumulative urinary excretion at steady state
Time Frame: Baseline and Day 30
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 16 | 14 | 14 | 22
mg | 1.72 (1.15) | 11.7 (5.84) | 30.9 (17.0) | 60.3 (27.1)

13. Secondary Outcome: Percent of LNP023 Excreted Into Urine at Day 30
Description: Percent of drug excreted into the urine
Time Frame: Baseline and Day 30
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Mean (Standard Deviation); unit: percent of dose
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 16 | 14 | 14 | 22
percent of dose | 8.59 (5.77) | 11.7 (5.84) | 15.5 (8.50) | 15.1 (6.77)

14. Secondary Outcome: Renal Clearance From Plasma at Steady State (CLr,ss) at Day 30
Description: The renal clearance from plasma at steady state
Time Frame: Baseline and Day 30
Population: PK analyses set - number of participants with evaluable results for each parameter
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID
Number analyzed (Participants) | 16 | 14 | 14 | 22
L/hr | 0.112 (0.0744) | 0.348 (0.179) | 0.719 (0.479) | 0.942 (0.540)

15. Secondary Outcome: Change From Baseline in Plasma Levels of Circulating Fragment of Factor B (Bb) and Soluble Terminal Complement Complex (sC5b-9) Biomarkers for Parts 1 and 2 to Day 90
Description: The complement AP biomarkers Bb and sC5b-9 were evaluated as potential pharmacodynamics and mode-of-action markers. Both biomarkers were measured using validated enzyme-linked immunosorbent assays (ELISAs).
Time Frame: Baseline, Days 8, 15, 30, 60, 90
Population: Full analysis set - all randomized patients with with a baseline and at least one post-baseline value
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 20 | 19 | 22 | 26 | 25
ng/mL
  Day 8 - Bb, n=14,16,13,25,19: number analyzed (Participants) | 14 | 16 | 13 | 25 | 19
  Day 8 - Bb, n=14,16,13,25,19 | 76.7 (22.89) | 72.2 (22.86) | 71.4 (30.66) | 66.3 (28.15) | 102.7 (19.78)
  Day 15 - Bb, n=13,14,16,22,22: number analyzed (Participants) | 13 | 14 | 16 | 22 | 22
  Day 15 - Bb, n=13,14,16,22,22 | 80.4 (32.59) | 74.1 (23.30) | 78.5 (33.35) | 72.9 (20.47) | 108.6 (23.19)
  Day 30 - Bb, n=16,17,18,26,24: number analyzed (Participants) | 16 | 17 | 18 | 26 | 24
  Day 30 - Bb, n=16,17,18,26,24 | 76.4 (18.32) | 76.2 (23.62) | 76.8 (34.00) | 70.4 (28.96) | 99.3 (22.07)
  Day 60 - Bb, n=14,16,17,25,21: number analyzed (Participants) | 14 | 16 | 17 | 25 | 21
  Day 60 - Bb, n=14,16,17,25,21 | 78.8 (20.26) | 75.2 (19.05) | 77.4 (35.23) | 72.8 (23.97) | 102.9 (24.07)
  Day 90 - Bb, n=17,16,17,25,21: number analyzed (Participants) | 17 | 16 | 17 | 25 | 21
  Day 90 - Bb, n=17,16,17,25,21 | 90.5 (25.57) | 79.3 (22.47) | 77.6 (35.42) | 74.6 (23.91) | 102.7 (22.01)
  Day 8 sC5B-9, n=12,16,13,22,17: number analyzed (Participants) | 12 | 16 | 13 | 22 | 17
  Day 8 sC5B-9, n=12,16,13,22,17 | 80.6 (12.29) | 69.6 (37.40) | 65.9 (24.05) | 75.8 (30.15) | 95.2 (22.01)
  Day 15 sC5B-9, n=13,14,16,21,21: number analyzed (Participants) | 13 | 14 | 16 | 21 | 21
  Day 15 sC5B-9, n=13,14,16,21,21 | 79.4 (27.60) | 72.2 (33.86) | 78.4 (33.35) | 78.0 (32.06) | 99.4 (25.40)
  Day 30 sC5B-9, n=16,17,18,25,24: number analyzed (Participants) | 16 | 17 | 18 | 25 | 24
  Day 30 sC5B-9, n=16,17,18,25,24 | 85.8 (23.88) | 68.6 (41.32) | 76.4 (25.97) | 69.8 (21.98) | 94.2 (24.96)
  Day 60 sC5B-9, n=14,16,17,24,20: number analyzed (Participants) | 14 | 16 | 17 | 24 | 20
  Day 60 sC5B-9, n=14,16,17,24,20 | 84.6 (27.37) | 73.7 (31.99) | 74.9 (29.65) | 76.2 (29.80) | 95.7 (30.11)
  Day 90 sC5B-9, n=16,16,17,23,19: number analyzed (Participants) | 16 | 16 | 17 | 23 | 19
  Day 90 sC5B-9, n=16,16,17,23,19 | 89.6 (28.66) | 73.8 (36.21) | 79.0 (22.82) | 75.0 (34.21) | 103.4 (21.52)

16. Secondary Outcome: Estimation of the Lowest Dose Providing Maximal Reduction of Proteinuria as Measured by the Ratio to Baseline in UPCR at Day 90
Description: The table shows the ratio to baseline in UPCR at Day 90 by treatment group. The lowest dose providing maximal reduction of proteinuria is the dose with the smallest UPCR ratio to baseline estimate (i.e. LNP023 200mg),
Time Frame: Baseline up to Month 3
Population: Full analysis set - all randomized patients with a baseline and at least one post-baseline value
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 22 | 26 | 25
Ratio to baseline | 0.85 [0.77 to 0.93] | 0.80 [0.73 to 0.87] | 0.76 [0.70 to 0.81] | 0.69 [0.61 to 0.77] | 0.88 [0.80 to 1.00]

17. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Change From Baseline for Estimated Glomerular Filtration Rate (eGFR) - Part 2 up to Day 180
Description: eGFR; estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Time Frame: Baseline and Day 180
Population: Full analysis set 2 - all randomized patients in study Part 2 that consented to receive treatment as per protocol version 04 or higher (i.e. 180 days of treatment)
Measure: Mean (Standard Error); unit: mL/min/SSA
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 9 | 10 | 19 | 11 | 11
mL/min/SSA | 0.78 (1.977) | -2.35 (1.995) | -2.91 (1.359) | -1.18 (1.798) | -3.17 (1.868)
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 3.95, 80% CI 2-sided [0.420 to 7.472]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 0.82, 80% CI 2-sided [-2.747 to 4.390]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Mean Difference (Final Values) = 0.26, 80% CI 2-sided [-2.745 to 3.262]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Mean Difference (Final Values) = 1.98, 80% CI 2-sided [-1.368 to 5.337]

18. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline Protein to Creatinine (UPCR) From 1st Morning Void - Part 2 up to Day 180
Description: A midstream urine sample was obtained from the first morning void (FMV) on the visit day.
Time Frame: Baseline and Day 180
Population: as for outcome 17
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 9 | 10 | 19 | 11 | 11
Ratio to baseline | 0.81 [0.599 to 1.108] | 0.72 [0.534 to 0.976] | 0.63 [0.507 to 0.784] | 0.72 [0.544 to 0.949] | 0.79 [0.590 to 1.047]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 1.04, 80% CI 2-sided [0.680 to 1.579]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.92, 80% CI 2-sided [0.607 to 1.390]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.80, 80% CI 2-sided [0.558 to 1.153]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.91, 80% CI 2-sided [0.614 to 1.362]

19. Secondary Outcome: Shift Table From Baseline for Hematuria Levels - Part 2 at Day 180
Description: Hematuria levels were the number of erythrocytes/high-power-field (hpf) measured through microscopic examination. The table shows the shift in hematuria grade (Low: <9 rbc/hpf, Intermediate: >=9 to <= 50 rbc/hpf, High: >50 rbc/hpf) from baseline (rows) to Day 180 (columns). A lower grade corresponds to a better outcome. Only patients with both baseline and Day 90 hematuria values are presented. L=low, I=intermediate and H=high in column headings for doses and BL=baseline
Time Frame: Baseline and Day 180
Population: Full analysis set - all randomized patients with both baseline and Day 180 hematuria values. The number of participants analyzed corresponds to the column totals (i.e. the number of patients with non-missing baseline and Day 180 values by hematuria level at Day 180 and treatment group).
Measure: Number; unit: participants
Groups:
- 10mg-L; 50mg-L; 100mg-L; 200mg-L; Pl-L: L (<9 rbc/hpf) at Day 180
- 10mg-I; 50mg-I; 100mg-I; 200mg-I; PL-I: I (>=9 to <= 50 rbc/hpf) at Day 180
- 10mg-H; 50mg-H; 100mg-H; 200mg-H; PL-H: H (>50 rbc/hpf) at Day 180
Arm/Group | 10mg-L | 10mg-I | 10mg-H | 50mg-L | 50mg-I | 50mg-H | 100mg-L | 100mg-I | 100mg-H | 200mg-L | 200mg-I | 200mg-H | Pl-L | PL-I | PL-H
Number analyzed (Participants) | 3 | 2 | 0 | 6 | 0 | 0 | 7 | 1 | 0 | 6 | 0 | 0 | 4 | 0 | 1
participants
  Low at baseline | 1 | 1 |  | 5 |  |  | 2 | 0 |  | 4 |  |  | 4 |  | 0
  Intermediate at baseline | 2 | 1 |  | 1 |  |  | 3 | 0 |  | 2 |  |  | 0 |  | 1
  High at baseline | 0 | 0 |  | 0 |  |  | 2 | 1 |  | 0 |  |  | 0 |  | 0

20. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Change From Baseline in Protein Level Urine Using the Urine Protein-creatinine Ratio (UPCR) From 24 Hour Urine Collection - Part 2 up to Day 180
Description: For UPCR test, participants collected all of their urine over a 24-hour period
Time Frame: Baseline, Days 30, 90 and 180
Population: as for outcome 17
Measure: Geometric Mean (80% Confidence Interval); unit: mg/d
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 9 | 10 | 19 | 11 | 11
mg/d | 1.06 [0.803 to 1.394] | 0.59 [0.452 to 0.779] | 0.66 [0.540 to 0.798] | 0.73 [0.568 to 0.940] | 0.91 [0.705 to 1.185]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Geometric mean ratio = 1.16, 80% CI 2-sided [0.792 to 1.692]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Geometric mean ratio = 0.65, 80% CI 2-sided [0.446 to 0.945]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Geometric mean ratio = 0.72, 80% CI 2-sided [0.518 to 0.997]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Geometric mean ratio = 0.80, 80% CI 2-sided [0.558 to 1.146]

21. Secondary Outcome: Mixed Model of Repeated Measures (MMRM) of the Ratio to Baseline in 24 Hour Urine Albumin to Creatinine (UACR) - Part 2 up to Day 180
Description: The 24-hour urine collection was started 1 day prior to the clinic visit, after participant urinated for the first time, than all urine was collected for the next 24 hours and refrigerated prior to clinic visit.
Time Frame: Baseline and Day 180
Population: as for outcome 17
Measure: Geometric Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LNP023 10 mg BID | LNP023 50 mg BID | LNP023 100 mg BID - Part 2 | LNP023 200 mg BID | Placebo
Number analyzed (Participants) | 9 | 10 | 19 | 11 | 11
Ratio to baseline | 1.04 [0.779 to 1.392] | 0.61 [0.454 to 0.808] | 0.65 [0.526 to 0.792] | 0.69 [0.533 to 0.902] | 0.91 [0.696 to 1.200]
Statistical Analysis 1: Comparison: LNP023 10 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 1.14, 80% CI 2-sided [0.765 to 1.699]
Statistical Analysis 2: Comparison: LNP023 50 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.66, 80% CI 2-sided [0.446 to 0.984]
Statistical Analysis 3: Comparison: LNP023 100 mg BID - Part 2 vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.71, 80% CI 2-sided [0.501 to 0.995]
Statistical Analysis 4: Comparison: LNP023 200 mg BID vs Placebo; Test type: Other; Ratio to placebo (of ratio to baseline) = 0.76, 80% CI 2-sided [0.520 to 1.107]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose to end of study treatment (tx) plus 7 days post tx. Maximum reporting time for Treatment Emergent Adverse Events was: Part 1=99 days, Part II: 197 days. There was an additional 90 day safety follow up period for both periods.
Groups:
- LNP023 10mg On-treatment: LNP023 10mg On-treatment
- LNP023 50mg On-treatment: LNP023 50mg On-treatment
- LNP023 100mg On-treatment: LNP023 100mg On-treatment
- LNP023 200mg On-treatment: LNP023 200mg On-treatment
- Placebo On-treatment: Placebo On-treatment
- LNP023 10mg Follow-up: LNP023 10mg safety follow-up
- LNP023 50mg Follow-up: LNP023 50mg follow-up
- LNP023 100mg Follow-up: LNP023 100mg follow-up
- LNP023 200mg Follow-up: LNP023 200mg follow-up
- Placebo Follow-up: Placebo follow-up
Arm/Group | LNP023 10mg On-treatment | LNP023 50mg On-treatment | LNP023 100mg On-treatment | LNP023 200mg On-treatment | Placebo On-treatment | LNP023 10mg Follow-up | LNP023 50mg Follow-up | LNP023 100mg Follow-up | LNP023 200mg Follow-up | Placebo Follow-up
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/22 | 0/26 | 0/25 | 0/20 | 0/19 | 0/22 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/19 | 0/22 | 0/26 | 1/25 | 1/20 | 1/19 | 2/22 | 1/26 | 1/25
Other Adverse Events (participants affected / at risk) | 14/20 | 16/19 | 15/22 | 14/26 | 17/25 | 6/20 | 5/19 | 5/22 | 10/26 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 10mg On-treatment (N=20) | LNP023 50mg On-treatment (N=19) | LNP023 100mg On-treatment (N=22) | LNP023 200mg On-treatment (N=26) | Placebo On-treatment (N=25) | LNP023 10mg Follow-up (N=20) | LNP023 50mg Follow-up (N=19) | LNP023 100mg Follow-up (N=22) | LNP023 200mg Follow-up (N=26) | Placebo Follow-up (N=25)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 10mg On-treatment (N=20) | LNP023 50mg On-treatment (N=19) | LNP023 100mg On-treatment (N=22) | LNP023 200mg On-treatment (N=26) | Placebo On-treatment (N=25) | LNP023 10mg Follow-up (N=20) | LNP023 50mg Follow-up (N=19) | LNP023 100mg Follow-up (N=22) | LNP023 200mg Follow-up (N=26) | Placebo Follow-up (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulation test abnormal (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystatin C increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test negative (Investigations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 1 | 3 | 1 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 2 | 6 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal vasculitis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03373461/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03373461/SAP_001.pdf